CLINICAL TRIAL: NCT01275742
Title: Testing a Brief Cognitive Therapy Intervention for Depressive Symptoms in Patients With Heart Failure
Brief Title: Helping Others Toward Positive Emotions in People With Heart Failure
Acronym: HOPE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rebecca L. Dekker, PhD, RN, APRN (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, Rebecca L. Dekker, PhD, RN, APRN, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5P20NR010679-04 (NIH); 5P20NR010679 (NIH)
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Heart Failure
Keywords: Heart failure; Depression; Depressive symptoms; Cognitive therapy; Hospitalization; Quality of life
MeSH Terms: conditions — Heart Failure; Depression | interventions — Cognitive Behavioral Therapy; Counseling; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Usual Care (No Intervention)
  Interventions: Behavioral: Brief Cognitive Therapy Intervention

INTERVENTIONS:
Behavioral: Brief Cognitive Therapy Intervention — The intervention group will receive an individual, 30 minute, scripted cognitive therapy session. This intervention will be delivered by an Advanced Practice Registered Nurse or a trained research nurse. An iPad will guide the outline of the intervention. The nurse will discuss depression in heart disease and the connection between thoughts, emotions, and behaviors. The nurse will ask the patient to describe a recent stressful experience and discuss thoughts that the patient has been experiencing. Two techniques for challenging negative thinking will be introduced to the patient: thought stopping and affirmations. The nurse will ask the patient to practice these techniques at home. After the patient has practiced both techniques, the nurse will leave the patient with a booklet with the intervention. At 1-2 weeks, the nurse will administer a booster session over the phone. This session will last 10-15 minutes and will reinforce the techniques learned during the brief CT intervention.
  Other Names: Cognitive therapy; Cognitive behavioral therapy; Counseling; Nursing intervention

SUMMARY:
Heart failure (HF) affects 5 million people in the US and is the most common cause of hospitalization in elderly adults. One-third of patients who are hospitalized with HF have major depression. Depressed HF patients have double the rates of morbidity and/or mortality and worse health-related quality of life than non-depressed HF patients. The investigators previous pilot research suggests that a brief Cognitive Therapy (CT) intervention may improve short-term cardiac survival among depressed hospitalized HF patients compared to non-depressed HF patients who received usual care. Therefore, the investigators will conduct a larger study to evaluate the effects of the intervention on longer cardiac event-free survival, symptoms of depression, health-related quality of life, and stress levels in patients with HF. The investigators hypothesize that patients in the intervention group will experience longer cardiac event-free survival, lower levels of depressive symptom, better health-related quality of life, and lower salivary cortisol levels at follow-up than patients who receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the hospital with a primary or secondary diagnosis of congestive heart failure OR admitted to the hospital for cardiac reasons and has a history of chronic heart failure
* American College of Cardiology/ American Heart Association Stage C HF
* 21 years or older

Exclusion Criteria:

* Co-existing terminal illness likely to be fatal within the next 12 months
* End-stage HF (defined as American College of Cardiology Stage D HF)
* Cognitive impairment that precludes the ability to give informed consent
* Active suicidality (defined choosing option 1, 2 or 3 on Item 9 of the PHQ-9)
* History of the death of a spouse or child within the past month
* History of psychotic illness or bipolar illness
* Current alcohol dependence or other substance abuse
* Non-English speaking or possessing any other communication barrier

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Cardiac event-free survival | Three months to five years
  To compare cardiac event-free survival at 3 months, 6 months, and up to five years between patients with HF and depressive symptoms who receive a brief cognitive therapy intervention (depressive symptom intervention group) and patients with HF and depressive symptoms who receive usual care (depressive symptom usual care group).

SECONDARY OUTCOMES:
Depressive symptoms | 1 week, 3 months, and 6 months
  Compare depressive symptoms at 1-week, 3 months, and 6 months between patients with HF and depressive symptoms who receive a brief CT intervention (depressive symptom intervention group) and patients with HF and depressive symptoms who receive usual care (depressive symptom usual care group).
Health-related quality of life | 1 week, 3 months, and 6 months
  Compare health-related quality of life at 1-week, 3 months, and 6 months between patients with HF and depressive symptoms who receive a brief CT intervention (depressive symptom intervention group) and patients with HF and depressive symptoms who receive usual care (depressive symptom usual care group).
Salivary cortisol | 1 week, 3 months, and 6 months
  Compare salivary cortisol at 1-week, 3 months, and 6 months between patients with HF and depressive symptoms who receive a brief CT intervention (depressive symptom intervention group) and patients with HF and depressive symptoms who receive usual care (depressive symptom usual care group).
No depressive symptom comparison group | 1 week, 3 months, and 6 months
  Compare cardiac event-free survival, depressive symptoms, health-related quality of life, and salivary cortisol levels between the depressive symptom intervention group and patients with HF and no depressive symptoms who receive usual care (no depressive symptom group) at 1-week, 3 months, and 6 months.
Salivary vs. serum biomarkers | Baseline
  Compare levels of salivary cortisol, BNP, CRP and IL-6 at baseline between patients with and without depressive symptoms, and determine whether the salivary measures of BNP, CRP, and IL-6 are correlated with serum measurement of these biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Dekker, PhD, Principal Investigator — University of Kentucky College of Nursing; Elizabeth Tovar, PhD, Principal Investigator — University of Kentucky College of Nursing
Locations (1):
- University of Kentucky Chandler Medical Center, Lexington, Kentucky, United States